CLINICAL TRIAL: NCT02110771
Title: Efficacy Study of GAÏA Program Cognitive Remediation of Facial Affects Processing in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Collaborators: Hospital Center Alpes-Isère (Other); Centre Hospitalier St Anne (Other); Centre Hospitalier Intercommunal Clermont de l'Oise (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-A00793-38
Record Dates: First submitted 2014-02-24; First posted 2014-04-10 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2015-09

CONDITIONS: Schizophrenia
Keywords: schizophrenia; social cognition; facial affects recognition; cognitive remediation
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GAÏA - facial affect recognition targeted (Experimental): GAÏA:20hours individual cognitive remediation with therapist, 10 tasks at home, 10 week-treatment cognitive remediation targeted on facial affects recognition. exercises were designed by Gaudelus and Franck (2012) and tutoractiv'company. It includes photos, computer and role games exercises.Computer based exercises have 5 difficulty levels.
  2 sessions of one hour per week with therapist.
  Tasks at home are given once a week and targeting functional outcomes associated with facial affects recognition impairment.
  Interventions: Behavioral: GAÏA - facial affect recognition targeted
- RECOS - attentional process targeted (Active Comparator): RECOS (Cognitive REmediation for Schizophrenia): 20 hours individual cognitive remediation with therapist, 10 tasks at home, 10 week-treatment.
  RECOS is a validated cognitive remediation program, developed by P. Vianin and SBT company. It includes paper and pen and computer based exercises. The original program proposes 5 modules targeting 5 cognitive functions, each patient participated in the module corresponding to his/her most altered cognitive function. In this study, all patients randomized in this arm are allocated in the attentional module.Every computer exercises have 10 difficulty levels.
  2 sessions of one hour per week with therapist.
  Tasks at home are given once a week and targeting functional outcome
  Interventions: Behavioral: RECOS - attentional process targeted

INTERVENTIONS:
Behavioral: GAÏA - facial affect recognition targeted — 2 sessions of one hour per week with therapist. Intervention proposes 3 stages : 1)discovering and learning facial affects recognition and discrimination criterions for joy, sadness and anger (photos exercises); 2) facial affect recognition training (computer based and role game exercises); 3) generalization to other emotions (photos, role games and computer based exercises).
  The therapist chooses the change of stages; 5 sessions or more are proposed for the generalization stage.
  Arms: GAÏA - facial affect recognition targeted
Behavioral: RECOS - attentional process targeted — 2 sessions of one hour per week with therapist the first of those two session is allocated to paper and pen exercises (search and validation of strategies to resolve cognitive training exercises or functional problems). the second session is allocated to computer based exercises.
  Arms: RECOS - attentional process targeted

SUMMARY:
Social cognition impairments was highlighted for persons suffering with schizophrenia by numerous studies. The use of treatment programs intended to treat specifically these deficits through procedures of cognitive remediation, will allow decreasing their impact on everyday life by improving abilities to understand and interact with others. Such tools could allow also profits in terms of reduction of positive and negative of schizophrenia. The Gaïa program is intended to improve the perception of the facial affects which is one of social cognition processes impaired in schizophrenia.

Methods:

This is a multicenter, randomized, controlled study comparing people aged 18 to 45 years with a diagnostic of schizophrenia according to the Diagnostic and Statistical manuel of Mental disorders, 4th edition (DSM-IV-TR).

The GAÏA program will be compared to an already validated neurocognitive remediation program, training attentional processes (RECOS).

100 patients will be randomized as follows: Arm 1, experimental: Gaïa (20h with therapist, computer assisted method) Arm 2, control: RECOS (20h with therapist, computer assisted method)

Condition: Schizophrenia Intervention: Behavioural: computer assisted cognitive remediation

Hypothesis:

A targeted cognitive remediation will more increased abilities in facial affects recognition processes than a non specific, attentional cognitive remediation.

Primary outcome measures:

- Change from baseline in performances in the Facial Emotion Recognition Task (TREF) after 10 weeks and 20 session of treatment.

Secondary outcome measures

* Change from baseline in clinical, psychosocial, social cognition and neurocognitive measures, after 10 weeks and 20 session of treatment and at 6 months follow-up.
* Change from baseline in performances in the Facial Emotion Recognition Task (TREF) after treatment and 6 months follow-up.

DETAILED DESCRIPTION:
Purpose:

Rationale:

Social cognition impairments was highlighted for persons suffering with schizophrenia by numerous studies. The use of treatment programs intended to treat specifically these deficits through procedures of cognitive remediation, will allow decreasing their impact on everyday life by improving abilities to understand and interact with others. Such tools could allow also profits in terms of reduction of positive and negative of schizophrenia. The Gaïa program is intended to improve the perception of the facial affects which is one of social cognition processes impaired in schizophrenia.

Methods:

This is a multicenter, randomized, controlled study comparing people aged 18 to 45 years with a diagnostic of schizophrenia according to the DSM-IV-TR.

The Gaïa program will be compared to an already validated neurocognitive remediation program, training attentional processes (RECOS).

100 patients will be randomized as follows:

1. Arm 1,Experimental: Gaïa (20h with therapist, computer assisted method)

   * 10 week-treatment, with 2 sessions of 1 hour per week, and 1 homework exercise without therapist per week.Individual therapy.
   * Gaïa exercises were designed by B. Gaudelus and tutoractiv' company, for specific use in schizophrenia. It includes computer based and paper & pen, photos and role games exercises targeting the recognition of facial emotions.
   * Computer based exercises have 5 increasing difficulty levels.
   * Each participant practices all the modules of Gaïa.
2. Arm 2, control: RECOS (20h with therapist, computer assisted method)

   * 10 week-treatment, with 2 sessions of 1 hour per week and 1 homework exercise without therapist per week.Individual therapy.
   * RECOS (Cognitive Remediation for Schizophrenia) exercises were designed by Scientific Brain Training (SBT) company and P. Vianin in year 2007 for specific use in schizophrenia.
   * It includes computer based and paper & pen exercises.
   * Only the RECOS attentional function module is used in the study (5 modules available in the program) with gradual difficulty in 10 levels

Condition: Schizophrenia Intervention: Behavioural: computer assisted cognitive remediation

Study type: interventional

Study design:

* Allocation: randomized
* Endpoint classification: efficacy study
* Intervention model: parallel assignment
* Masking: Single Blind (outcomes assessor)
* Primary purpose: treatment

Official title:

Efficacy study of GAÏA program; cognitive remediation of facial affects process in schizophrenia

Hypothesis:

A targeted cognitive remediation will more increased abilities in facial affects recognition processes than a non specific, attentional cognitive remediation.

Primary outcome measures:

- Change from baseline in performances in the Facial Emotion Recognition Task (TREF) after 10 weeks and 20 session of treatment.

Secondary outcome measures

* Change from baseline in clinical and psychosocial measures, including symptoms, Delusional ideas, self esteem, insight and functional outcome after 10 weeks and 20 session of treatment and at 6 months follow-up.
* Change from baseline in social cognition measures, including Theory of Mind,attribution style, emotional conciousness and empathy processes after 10 weeks and 20 session of treatment and at 6 months follow-up
* Change from baseline in neurocognitive functioning measures, including attentional, working memory, processing speed, perceptive and executive functions processes after 10 weeks and 20 session of treatment and at 6 months follow-up.
* Change from baseline in performances in the Facial Emotion Recognition Task (TREF) after treatment and 6 months follow-up.

  1. Scales for clinical and psychosocial functioning measurement:
* Positive and negative symptoms scale (PANSS)
* Peters and al. Delusions Inventory 21 items (PDI21)
* Birchwood insight scale
* Self-Esteem Rating Scale (SERS)
* Social Autonomy Scale (EAS)

  2. Tasks for social cognitive measurement
* Hinting task - Theory of mind
* Intentional Reading in Situation - Theory of mind - (LIS-V)
* Eyes Test - Theory of mind
* Ambiguous Intentions Hostility Questionary - Attribution style - (AIHQ)
* Levels of Emotional Awareness Scale (LEAS)
* Questionnaire of Cognitive and Affective Empathy (QCAE)

  3. Tasks for neurocognitive functioning measurement
* Attentional functions: D2 test ; Attentional Testbattery (TAP)
* Executive functions: Trail making test (TMT); Search keys score - Behavioural Assessment of Dysexecutive functions (BADS); Rey figure
* Working memory: memory span ; Corsi blocs ; Brief Visual Memory Test- Revised (BVMT-R) processing speed: Wechsler Adult Intelligence Scale IV - Code and Symbol score (WAIS IV) perceptive functions: HOOPER Visual Organization Test (VOT)

Eligibility

* Ages Eligible for Study: 18 years to 45 years
* Genders Eligible for Study: Both
* Accepts Healthy volunteers: No

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 45 years
* French speaker
* Clinical stability
* Diagnosis of schizophrenia according to the DSM-IV-TR
* Agreement of the guardian for the patients under guardianship
* Unchanged psychotropic treatment during month preceding the inclusion
* Overdrawn performances in the treatment of the facial information
* Patients having given their consent lit to participate in the study

Exclusion Criteria:

* alcohol or drug dependence (according to the DSM-IV-TR), except tobacco
* history of neurobiological illness or trauma
* the ineffectiveness of neuroleptic treatment
* Taking of medicine with somatic aim having a cerebral or psychic impact
* Simultaneous participation on an other program of cognitive remediation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2012-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Facial Emotions Recognition Task(TREF) | week 11
  The TREF presents 54 photos representing 6 basic emotions (joy, anger, sadness, fear, disgust and contempt). Each emotion is presented with 9 intensity levels (from 20% to 100%),and by 4 models (2 mens and 2 womens) Subject has to select his answer in a list of 6 items (joy, anger, sadness, fear, disgust and contempt), each photo is presented during 10 seconds maximum, there's no time limit to answer.

SECONDARY OUTCOMES:
TREF (Facial emotions recognition task) | 6 month follow up
Change from baseline in symptoms measure 1 | week 11 and 6 month follow-up
  PANSS - Positive and negative symptoms scale. global score, positive sub scale score and negative sub scale score
Change from baseline in social cognition measures | week 11 and 6 month follow-up
  Tasks for social cognitive measurement: Hinting task - Theory of mind ; LIS-V - Theory of mind - intentional reading in situation; Eyes Test - Theory of mind ; AIHQ- Attribution Style ; Ambiguous Intentions Hostility Questionary ; LEAS- Levels of Emotional Awareness Scale; QCAE- Questionnaire of Cognitive and Affective Empathy
Change from baseline in neurocognitive functioning measures | week 11and 6 month follow-up
  Tasks for neurocognitive functioning measurement attentional functions: D2; TAP. Executive functions:TMT- Trail making test ; BADS/search keys score ; Rey figure. Working memory: memory span ; Corsi blocs ;BVMT-R. Processing speed: WAIS-IV - Code and Symbol score. Perceptive functions: VOT.
Change from baseline in symptoms measure 2 | week 11 and 6 month follow-up
  PDI 21- Peters and al. Delusions Inventory 21 items Global score
Change from baseline in insight measure | week 11 and 6 month follow-up
  Birchwood insight scale. Global score
Change from baseline in self estime measure | week 11 and 6 month follow up
  SERS -Self-Esteem Rating Scale. Global score
Change from baseline in social functioning measure | week 11 and 6 month follow-up
  EAS -Social Autonomy Scale. Global score and relationship with others score

CONTACTS AND LOCATIONS:
Overall Officials: Franck Nicolas, PUPH, Principal Investigator — Hôpital le Vinatier
Locations (1):
- centre de réhabilitation - Hôpital le Vinatier, Lyon, Rhône, France

REFERENCES:
- [Background] Vianin P.Cognitive Remediation for schizophrenia. Presentation of the RECOS program.Anales Medico psychologiques 165: 200-205, 2007
- [Background] Franck N, Duboc C, Sundby C, Amado I, Wykes T, Demily C, Launay C, Le Roy V, Bloch P, Willard D, Todd A, Petitjean F, Foullu S, Briant P, Grillon ML, Deppen P, Verdoux H, Bralet MC, Januel D, Riche B, Roy P; Other members of the Cognitive Remediation Network; Vianin P. Specific vs general cognitive remediation for executive functioning in schizophrenia: a multicenter randomized trial. Schizophr Res. 2013 Jun;147(1):68-74. doi: 10.1016/j.schres.2013.03.009. Epub 2013 Apr 9. PMID 23583327
- [Background] Gaudelus B, Franck N. Troubles du traitement des informations faciales. Le programme GAÏA. In Franck N, editor.La remédiation cognitive. Paris: Eselvier Masson: 169-81,2012.
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Peters E, Joseph S, Day S, Garety P. Measuring delusional ideation: the 21-item Peters et al. Delusions Inventory (PDI). Schizophr Bull. 2004;30(4):1005-22. doi: 10.1093/oxfordjournals.schbul.a007116. PMID 15954204
- [Background] Birchwood M, Smith J, Drury V, Healy J, Macmillan F, Slade M. A self-report Insight Scale for psychosis: reliability, validity and sensitivity to change. Acta Psychiatr Scand. 1994 Jan;89(1):62-7. doi: 10.1111/j.1600-0447.1994.tb01487.x. PMID 7908156
- [Background] Lecomte T, Corbiere M, Laisne F. Investigating self-esteem in individuals with schizophrenia: relevance of the Self-Esteem Rating Scale-Short Form. Psychiatry Res. 2006 Jun 30;143(1):99-108. doi: 10.1016/j.psychres.2005.08.019. Epub 2006 May 24. PMID 16725210
- [Background] Leguay D, Cochet A, Matignon G, Hairy A, Fortassin O, Marion JM. [Social Autonomy Scale. First validation data]. Encephale. 1998 Mar-Apr;24(2):108-19. French. PMID 9622789
- [Background] Corcoran R, Frith CD. Thematic reasoning and theory of mind. Accounting for social inference difficulties in schizophrenia. Evolutionary Psychology 3, 2005.
- [Background] Bazin N, Brunet-Gouet E, Bourdet C, Kayser N, Falissard B, Hardy-Bayle MC, Passerieux C. Quantitative assessment of attribution of intentions to others in schizophrenia using an ecological video-based task: a comparison with manic and depressed patients. Psychiatry Res. 2009 May 15;167(1-2):28-35. doi: 10.1016/j.psychres.2007.12.010. Epub 2009 Apr 5. PMID 19346006
- [Background] Baron-Cohen S, Wheelwright S, Hill J, Raste Y, Plumb I. The "Reading the Mind in the Eyes" Test revised version: a study with normal adults, and adults with Asperger syndrome or high-functioning autism. J Child Psychol Psychiatry. 2001 Feb;42(2):241-51. PMID 11280420
- [Background] Combs DR, Penn DL, Wicher M, Waldheter E. The Ambiguous Intentions Hostility Questionnaire (AIHQ): a new measure for evaluating hostile social-cognitive biases in paranoia. Cogn Neuropsychiatry. 2007 Mar;12(2):128-43. doi: 10.1080/13546800600787854. PMID 17453895
- [Background] Reniers RL, Corcoran R, Drake R, Shryane NM, Vollm BA. The QCAE: a Questionnaire of Cognitive and Affective Empathy. J Pers Assess. 2011 Jan;93(1):84-95. doi: 10.1080/00223891.2010.528484. PMID 21184334
- [Background] Bydlowski S, Corcos M, Paterniti S, Guilbaud O, Jeammet P, Consoli SM. [French validation study of the levels of emotional awareness scale]. Encephale. 2002 Jul-Aug;28(4):310-20. French. PMID 12232540
- [Background] Gaudelus B, Virgile J, Peyroux E, Leleu A, Baudouin JY, Franck N. [Measuring impairment of facial affects recognition in schizophrenia. Preliminary study of the facial emotions recognition task (TREF)]. Encephale. 2015 Jun;41(3):251-9. doi: 10.1016/j.encep.2014.08.013. Epub 2014 Sep 17. French. PMID 25240938